CLINICAL TRIAL: NCT02358395
Title: A Phase I Study of BBI608 Administrated With Sorafenib in Adult Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Study of BBI608 Administrated With Sorafenib in Adult Patients With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8808001
Record Dates: First submitted 2015-01-21; First posted 2015-02-09 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — napabucasin; Sorafenib

ARMS (1):
- BBI608 puls Sorafenib (Experimental)
  Interventions: Drug: BBI608; Drug: Sorafenib

INTERVENTIONS:
Drug: BBI608 — Administered continuously twice daily with doses separated by 9-15 hours.
Drug: Sorafenib — Sorafenib 400 mg twice daily (800 mg total daily dose).

SUMMARY:
This is an open-label, multicenter, phase 1 study of BBI608 in combination with Sorafenib. This study population is adult Japanese patients with advanced hepatocellular carcinoma in Sorafenib combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or diagnosed imaging with hepatocellular carcinoma, and not indicated with a)-d) .

  1. Radiofrequency ablation therapy (RFA)
  2. Local therapy [such as percutaneous transhepatic ethanol injection therapy (PEIT), Microwave coagulation therapy (MCT)]
  3. Transcatheter arterial embolization (TAE)
  4. Transcatheter arterial chemoembolization (TACE)
* ≥ 20 years of age.
* Not treatment with systemic chemotherapy.
* Signed written informed consent must be obtained and documented.
* Life expectancy ≥ 3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Must be Child Pugh Class A.
* Hemoglobin ≥ 8.5 mg/dl.
* Absolute neutrophil count ≥ 1.5 x 10^9 /L.
* Platelets ≥ 75 x 10^9/L.
* Creatinine ≤ 1.5 x ULN.
* Total Bilirubin ≤ 3.0 mg/dl.
* Aspartate Aminotransferase (AST) and Alanine transaminase (ALT) ≤ 5.0 x the upper limit of normal (ULN).
* Females of childbearing potential must have a negative serum pregnancy test.
* Male or female patients of child-producing potential must agree to use contraception or avoidance of pregnancy measures during the study and for 30 days after the last BBI608 dose.

Exclusion Criteria:

* Have had any t a)-i) treatment less than 28 days prior to beginning the enrolment.

  1. Radiation therapy
  2. Hormone therapy
  3. Immune therapy
  4. Hyperthermia
  5. Surgical procedure
  6. Local therapy (such as RFA, PEIT, MCT)
  7. TAE
  8. TACE
  9. other anti- tumour treatment
* Have had a brain metastases with a symptom or requiring treatment.
* Have had coinstantaneous active multiple cancers.
* Have had a carcinomatous pleural effusion, ascites, or cardiac effusion requiring treatment.
* Esophageal varix requiring treatment.
* Patient of pregnancy or possibility of pregnancy, and planning breastfeeding by the end of BBI608 administration after 30days.
* Crohns disease, ulcerative colitis, or historical surgery of extensively small intestine resection.
* Unable or unwilling to swallow BBI608 capsules or Sorafenib tablets.
* Uncontrolled inter-current illness (such as Grade 3active infection, or serious respiratory disease).
* HIV infection.
* Abnormal ECGs which are clinically significant within 28 days before enrolment.
* Patients who are New York Heart Association (NYHA) functional classes III, or IV, or unstable angina.
* Patients newly expressing angina within three months before the enrolment.
* Have had myocardial infarction within six months before the enrolment.
* Administrating with antiarrhythmic drug.
* Have received other investigational products or post-marketing investigational products within 4 weeks of the first dose of BBI608.
* Prior treatment with BBI608.
* Hypersensitivity to Sorafenib or any other component of Sorafenib.
* Ineligible for participation in the study in the opinion of the Investigators.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Assessment of safety and tolerability of BBI608 given in combination with Sorafenib by reporting of adverse events and serious adverse events. | 7 month
Assessment of dose-limiting toxicities (DLTs). | 29 days
Pharmacokinetic profile of BBI608 when administered in combination with Sorafenib. | On day 1: Prior to BBI608 dosing and 2,4,6,8,10,12 and 24 hours after the first dose. On day 29: Prior to BBI608 dosing and 2,4,6,8,10,12 and 24 hours after the first dose.

SECONDARY OUTCOMES:
Assessment of the preliminary anti-tumour activity. | Approximately 7 months
  Anti-tumour activity is assessed every 8 weeks from the first dose of BBI608 after the last dose of BBI608.The radiologic assessments will be evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and modified RECIST for patients with hepatocellular carcinoma.
Progression Free Survival | Approximately 7 month
  The time the participant stays on study until progression will be measured and recorded.
Overall Survival | Approximately 1 year
  Participants follow-up for overall survival will occur. Maximum follow-up time is 1 year after the initial administration of the last subject.

CONTACTS AND LOCATIONS:
Overall Officials: Director, Drug Development Division, Study Director — Sumitomo Pharma Co., Ltd.
Locations (1):
- 4 Sites, Tokyo,etc, Japan

REFERENCES:
- [Derived] Okusaka T, Morimoto M, Eguchi Y, Nakamura S, Iino S, Kageyama R. A Phase I Study to Investigate the Safety, Tolerability and Pharmacokinetics of Napabucasin Combined with Sorafenib in Japanese Patients with Unresectable Hepatocellular Carcinoma. Drugs R D. 2023 Jun;23(2):99-107. doi: 10.1007/s40268-023-00416-8. Epub 2023 May 15. PMID 37188895